CLINICAL TRIAL: NCT02872675
Title: The Effects of HOST-DM059 Prebiotic Supplementation on Gut Bacterial Metabolites, and Markers of Systemic Inflammation in Adults With and Without Hyperpnoea-Induced Bronchoconstriction: A Double-Blind, Placebo-Controlled, Crossover Trial.
Brief Title: The Effects of Prebiotics on Gut Bacterial Parameters, Immune Function & Exercise-Induced Airway Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: University of Reading (Other); Clasado Biosciences (Unknown); Imperial College London (Other); HOST Therabiomics (Unknown); The John van Geest Cancer Research Centre (Unknown)
Responsible Party: Principal Investigator, Paul Lester, PhD Student, Principal Investigator, Nottingham Trent University
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 233556
Record Dates: First submitted 2016-08-04; First posted 2016-08-19 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Exercised Induced Asthma; Asthma
Keywords: Asthma; Exercise-Induced Asthma; Gut Bacteria; Bimuno® Galactooligosaccharide; Pulmonary Function; Prebiotics; Exercise-Induced Bronchoconstriction; Gut Microbiota; Nutritional Intervention; Eucapnic Voluntary Hyperpnoea; Systemic Inflammation; Systemic Immune Function; Regulatory T Cells; TH1 Cells; TH2 Cells; Short-Chain Fatty Acids; Acetate; Propionate; Butyrate; Metabolomics; Airway Inflammation; Intestinal Permeability
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma | interventions — Prebiotics; maltodextrin

STUDY DESIGN:
Intervention Model Description: Participants will be administered a prebiotic (galactooligosaccharide; HOST-DM059), and a taste/appearance matched placebo (Maltodextrin) in a, double-blind, placebo-controlled, crossover design.
  The nutritional intervention will be completed over a twelve week period, consisting of two, four-week supplementation phases separated by a four-week wash out period. Participants will be randomly allocated one of the nutritional supplements during phase one (labelled as either 'L', or 'X'), and asked to consume one powdered sachet every morning (3.6g). Participants will then complete a four week wash out period, before being assigned the remaining nutritional supplement during phase two. Sachets can be reconstituted in tea/coffee/fruit juice, or sprinkled over cereal etc.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the company providing the nutritional supplements (HOST Therabiomics) will be aware of the supplement blinding protocol.
  Upon trial completion (e.g. the final visit of the final participant), the chief investigator will contact HOST Therabiomics to obtain information on the supplement blinding protocol. Should any participants, care providers, investigators, or outcome assessors become aware of the blinding protocol during the trial they will be informed not to disclose this information to any other relevant personnel. Participants who become aware of the blinding protocol during participation would be withdrawn from the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOST-DM059 (Prebiotic) (Experimental): HOST-DM059 is the only Second Generation Prebiotic, manufactured by Clasado Biosciences/HOST Therabiomics. HOST-DM059 consists of a specific type of carbohydrate/dietary fibre (GOS), and an enzyme extracted from species of Bifidobacteria (e.g. The β-Galacotosidase Enzyme, & Bifidobacterium Bifidum). The enzyme from which HOST-DM059 is developed provides a highly selective source of energy for certain species of Bifidobacteria. HOST-DM059 encourages the growth and development of Bifidobacteria. Certain species of Bifidobacteria have been demonstrated to exert prominent immunomodulatory effects in terms of regulating systemic inflammation.
  Interventions: Dietary Supplement: HOST-DM059
- Maltodextrin (Placebo Comparator): Maltodextrin will be administered as a taste/appearance-matched sugar/carbohydrate.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: HOST-DM059 — Experimental Supplement: HOST-DM059.
  Participants will be asked to orally consume one powdered sachet each day, at the same time in the morning, reconstituted in tea/coffee/fruit juice, or sprinkled over cereal etc. Whichever method of consumption is chosen, this must be kept consistent across both supplementation phases.
  Other Names: Bimuno, B-GOS, Prebiotic, Galactooligosaccharide.
  Arms: HOST-DM059 (Prebiotic)
Dietary Supplement: Maltodextrin — Placebo Comparator: Maltodextrin.
  Other Names: Placebo
  Arms: Maltodextrin

SUMMARY:
The current study aims to explore the role of prebiotic supplementation in adults with and without Asthma/Exercise-Induced Bronchoconstriction (A/EIB). All participants will be asked to consume a prebiotic supplement, and a placebo, each for a total duration of four weeks, separated by a two-week wash out period. The investigators hypothesise that improvements in pulmonary function observed in adults with Asthma following prebiotic supplementation. We hypothesise that improvements in pulmonary function will be attributed, at least in part, to gut microbiota mediated improvements in human immune function.

DETAILED DESCRIPTION:
The current study will investigate the effects of prebiotic supplementation on airway inflammation/bronchoconstriction in adults diagnosed with Asthma/Exercise-Induced Bronchoconstriction (A/EIB). Previous research conducted in adults diagnosed with A/EIB has reported significant improvements in pulmonary function following three weeks of prebiotic supplementation. The significant improvements in pulmonary function were attributed to an attenuation of various markers of airway inflammation, potentially regulated by gut microbiota mediated improvements in systemic immune function.

Prebiotics are a type of non-digestible carbohydrate/dietary fibre that can only be digested by certain beneficial bacteria. During the fermentation of prebiotics, beneficial bacteria produce energy/metabolites that can be used to support a variety of human immune functions, such as reducing the level of airway inflammation that occurs following exposure to relevant triggers (e.g. exercise).

Imbalances and/or deficiencies in gut bacterial composition/metabolic activity have been identified in children/adults diagnosed asthma. However, the potential mechanisms behind prebiotic mediated improvements in the severity of asthma have yet to be investigated.

Participants with and without A/EIB will be allocated two separate nutritional supplements following a double-blind, placebo-controlled design. During the first phase of the nutritional intervention, participants will consume the first supplement (either prebiotic or placebo), for a total duration of four weeks. A two-week wash out period will then be completed before the remaining nutritional supplement is administered for an equal duration.

Analyses of key human/bacterial metabolite concentrations will be carried out alongside assessments of immune and pulmonary function, and intestinal permeability at baseline, and throughout all phases of the nutritional intervention. Current understandings of the role of the gut microbiota in the pathogenesis of A/EIB will be expanded through the investigation of novel pathophysiological mechanisms, helping to inform future therapeutic prospects for asthma.

ELIGIBILITY:
Inclusion Criteria:

Be 18-50 years of age at the date of your first visit.

Have a body mass index (BMI) of 18.5-25 kg∙m2 (this will be worked out by the researchers using the participant's height and body weight).

Be physically active (completing 3 or more exercise sessions a week lasting at least 45 minutes each).

Be a non-smoker.

Asthma is defined as Steps 1, 2, or 3 based on British Thoracic Society guidelines.

Asthma sufferers must have a current medication prescription from their GP (e.g. maintenance/reliever inhalers).

In the researcher's opinion, the participant is able and willing to follow all trial requirements.

Exclusion Criteria

Asthma defined as Steps 4 or 5 based on British Thoracic Society guidelines.

Asthma sufferers who do not have a current medication prescription from their GP (e.g. maintenance and reliever inhalers).

Regular consumption of Omega-3 supplements, and/or high levels of Omega-3 intake from food (e.g. consuming more than 1-2 portions of oily fish such as salmon or mackerel a week).

Regularly consume antioxidant supplements.

Standard multivitamin and mineral supplements are acceptable, as long as the product label states the recommended Dietary Reference Values (DRV's).

If a single antioxidant supplement (e.g. Vitamin C), exceeds the recommended daily DRV's this will be checked with the chief investigator.

Take a daily dose of aspirin or other non-steroidal anti-inflammatory drugs such as ibuprofen.

Have consumed prebiotics and/or probiotics, drugs that affect gastrointestinal mobility, or laxatives in the 4 weeks before participation.

Currently taking a daily dose of anti-histamine, which could not be refrained from for 72 hours before each testing session.

Unable to refrain from taking Asthma medication (e.g. maintenance and reliever inhalers) for a prescribed duration before each testing session (e.g. 8-96 hours).

Vegetarian or vegan diet.

Previously diagnosed with chronic obstructive pulmonary disease (COPD), emphysema, chronic bronchitis, or similar respiratory illness.

Participants with asthma that have ever been hospitalised due to asthma (e.g. intensive care unit).

Participants with asthma that have received treatment with oral corticosteroids/been admitted to hospital during the past 12 months for their asthma.

An increase/step-up in asthma medication during the study (e.g. moving from Step 1 to Step 2, Step 2 to Step 3 etc.).

Participants with asthma who do not obtain an additional prescription for a reliever inhaler to be stored securely at NTU if needed during visits. Additional prescriptions must be obtained before familiarisation/visit two. Participants will be reimbursed for the cost of additional reliever inhaler prescriptions.

History of heart failure, pulmonary hypertension, embolism, or other pulmonary heart disease.

History of recurrent chest infections.

Smoker.

Pregnant, planning pregnancy or lactating.

Had an acute infection in the last four weeks, and/or major operation in the past four months.

History of gastrointestinal drug reaction.

Have taken antibiotics in the past 3 months.

History or current evidence of gastrointestinal disease (e.g. chronic constipation, diarrhoea, irritable bowel syndrome, Chrohn's disease).

Have recently taken part in other research projects. Participants will be asked to notify the chief investigator.

Participants are, or believe that they are lactose intolerant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Changes In Regulatory T Cell FOXP3 Expression From Baseline To Post Prebiotic Supplementation. | Week 0, Week 4, Week 6, Week 10 (Collected At Rest).
  Flow Cytometric Analysis: CD4+ CD25+ IL-10+ Regulatory T Cell FOXP3 Expression (

SECONDARY OUTCOMES:
Change In Systemic Immune Function/Inflammatory Markers | Week 0, Week 4, Week 6, Week 10 (Blood Sample Collected At Rest).
  Flow Cytometric Analysis: Interleukin (IL)-10, Hematopoietic Prostaglandin D Synthase Enzyme (Pathogenic Effector/Non-Pathogenic Effector TH2 Cells), CD3 (T Cells), CD25 (Regulatory T Cells), Transforming Growth Factor-Beta (TH2 Cells), Fork-Head Box Protein-3 (Regulatory T Cells), CD161 (PETH2 Cells), Interferon-Gamma (TH1 Cells), Live/Dead, Total & Specific White Blood Cell Counts (Eosinophils, Basophils, Neutrophils, Monocytes, Lymphocytes).
Change In Pulmonary Function (FEV1) | Week 0, Week 4, Week 6, Week 10 (At Rest & In Duplicate At 3, 6, 10, 15, 20, & 30 Minutes Post EVH).
  % Drop In Pulmonary Function (FEV1) Post EVH = 100*(Highest Baseline FEV1-Lowest Post EVH FEV1)/Highest Baseline FEV1. Used To Objectively Diagnose Asthma/EIB (> 10% Drop In FEV1 Post EVH At Two Consecutive Time Points), And Classify Severity As Mild (> 10% - < 25% Drop In FEV1), Moderate (> 25% - < 50% Drop In FEV1), Or Severe (> 30%, Or 50% Drop In FEV1 For Patients Receiving/Not Receiving Steroid Based Treatments).
  All Pulmonary Function Parameters: FEV1, FVC, PEF, FEF25%-75%.
  > 10% Reduction = Positive Objective Diagnosis (Asthma/EIB).
Change In The Asthma Control Questionnaire - Perceived Symptom Management | Weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10. (Upon Experimental Trial Arrival During Weeks 0, 4, 6, & 10).
  Common Asthma Symptoms Management: Night Time Awakening, Upon Waking Symptom Severity, Physical Activity Limitation, Dyspnoea (Breathlessness), Wheezing, Reliever Medication Usage (Rating 0-6).
Change In Urinary Metabolite Concentrations | Week 0, Week 4, Week 6, Week 10 (Urine Sample) (Collected At Rest & 60 Minutes Post EVH).
  E.G.: Acetic Acid, Propionic Acid, I-Butyric Acid, N-Butyric Acid, I-Valeric Acid, N-Valeric Acid, N-Caproic Acid.
Change In The Medication Adherence Report Scale For Asthma (MARS-A) | Weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10. (Upon Experimental Trial Arrival During Weeks 0, 4, 6, & 10).
  Asthma Medication & Nutritional Interventions Adherence Measurement (12 Questions) (Rating 1-5).
Change In 24 Hour Weighed Nutritional Intake Record | Week 0, Week 4, Week 8, Week 12 (24 Hours Before Experimental Trial).
  Quantitative Measurement - Habitual Nutritional Consumption (Assess Nutritional Intake Consistency Across Experimental Trials).
Changes In Intestinal Permeability Markers | Week 0, Week 4, Week 6, Week 10 (Blood Sample Collected At Rest).
  Blood (Serum/Plasma) Based Measurement.

OTHER OUTCOMES:
Principal Component Analysis/Cluster Analysis - Primary/Secondary Outcome Measures | Post Data Collection.
  All Relevant Meta-Data.
Partial Least Squares Discriminant Analysis. | Post Data Collection.
  Urinary Metabolite Profiles.
  Untargetted Metabolomics.
  1H Nuclear Magnetic Resonance (NMR) Spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Graham R Sharpe, PhD, Study Director — Nottingham Trent University
Locations (1):
- Nottingham Trent University, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may be made available to other researchers following completion of the current trial in an anonymised/pseudonymised format to prevent individual participant identification. Data will be provided in response to certain requests (e.g. if a systematic review and meta-analysis/statistical power calculation is being conducted that requires access to certain raw data).

REFERENCES:
- [Background] Williams NC, Johnson MA, Hunter KA, Sharpe GR. Reproducibility of the bronchoconstrictive response to eucapnic voluntary hyperpnoea. Respir Med. 2015 Oct;109(10):1262-7. doi: 10.1016/j.rmed.2015.08.006. Epub 2015 Aug 13. PMID 26303339
- [Background] Vulevic J, Juric A, Walton GE, Claus SP, Tzortzis G, Toward RE, Gibson GR. Influence of galacto-oligosaccharide mixture (B-GOS) on gut microbiota, immune parameters and metabonomics in elderly persons. Br J Nutr. 2015 Aug 28;114(4):586-95. doi: 10.1017/S0007114515001889. Epub 2015 Jul 28. PMID 26218845
- [Background] Williams NC, Johnson MA, Shaw DE, Spendlove I, Vulevic J, Sharpe GR, Hunter KA. A prebiotic galactooligosaccharide mixture reduces severity of hyperpnoea-induced bronchoconstriction and markers of airway inflammation. Br J Nutr. 2016 Sep;116(5):798-804. doi: 10.1017/S0007114516002762. PMID 27523186
- [Background] Hevia A, Milani C, Lopez P, Donado CD, Cuervo A, Gonzalez S, Suarez A, Turroni F, Gueimonde M, Ventura M, Sanchez B, Margolles A. Allergic Patients with Long-Term Asthma Display Low Levels of Bifidobacterium adolescentis. PLoS One. 2016 Feb 3;11(2):e0147809. doi: 10.1371/journal.pone.0147809. eCollection 2016. PMID 26840903
- [Background] Arrieta MC, Stiemsma LT, Dimitriu PA, Thorson L, Russell S, Yurist-Doutsch S, Kuzeljevic B, Gold MJ, Britton HM, Lefebvre DL, Subbarao P, Mandhane P, Becker A, McNagny KM, Sears MR, Kollmann T; CHILD Study Investigators; Mohn WW, Turvey SE, Finlay BB. Early infancy microbial and metabolic alterations affect risk of childhood asthma. Sci Transl Med. 2015 Sep 30;7(307):307ra152. doi: 10.1126/scitranslmed.aab2271. PMID 26424567